CLINICAL TRIAL: NCT00882245
Title: A Phase II, Double-Blind, Vehicle Controlled Study to Determine the Efficacy, Safety and Toleration of SRD441 Ointment in Patients With Atopic Dermatitis
Brief Title: Safety and Efficacy of SRD441 Ointment in Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Serentis Ltd. (Industry)
Responsible Party: Robert Tansley, Chief Medical Officer, Serentis Ltd
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P441201CD
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2009-10-30 (Estimated); Status verified 2009-10

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Ointments

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vehicle ointment (Placebo Comparator)
  Interventions: Other: Vehicle ointment
- SRD441 Ointment (Experimental)
  Interventions: Drug: Ointment

INTERVENTIONS:
Other: Vehicle ointment — Topical vehicle cream
  Arms: Vehicle ointment
Drug: Ointment — SRD441 Ointment
  Arms: SRD441 Ointment

SUMMARY:
Atopic Dermatitis is a chronic inflammatory skin disease that affect 10 to 15% of children and 2 to 10% of adults. AD is characterised by an itchy skin eruption and may cover large parts of the body. The exact cause is unknown but is thought to be an interplay between genetic and and environmental factors. The objective of this study is to determine whether SRD441 ointment is a safe and effective therapy for mild to moderate Atopic Dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 or over
* Subjects with a history of AD
* Written and dated informed consent
* Satisfactory medical assessment with no clinical relevant abnormalities.

Exclusion Criteria:

* Subjects with current or recurrent disease (except AD) that could affect the site of application, the action, absorption or disposition of the investigational product, or clinical or laboratory assessments.
* Subjects who have medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgement of the investigator, would make the subject inappropriate for entry into this trial.
* Subjects with any skin tattoo, scar, cuts, bruises, or other skin damage, including excessive UV exposure, at the possible drug application sites which could impact the application of the test agent or confound the local assessments during this study.
* Subjects with clinically significant renal and liver parameters, as defined as greater than 1.5 x creatinine and 3 x AST ULN (upper limit of normal) respectively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2009-04; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Measure efficacy in treating acute exacerbations | 4 weeks

SECONDARY OUTCOMES:
Safety and local dermal tolerability | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert Tansley, Study Director — Serentis Ltd.
Locations (12):
- Bulgaria (2):
  - Plovdiv
  - Sofia
- Helsinki, Finland
- Germany (9):
  - Berlin
  - Bonn
  - Cologne
  - Frankfurt
  - Hanover
  - Heidelberg
  - Kiel
  - Munich
  - Münster

REFERENCES:
- [Derived] Foelster Holst R, Reitamo S, Yankova R, Worm M, Kadurina M, Thaci D, Bieber T, Tsankov N, Enk A, Luger T, Duffy M, Tansley R. The novel protease inhibitor SRD441 ointment is not effective in the treatment of adult subjects with atopic dermatitis: results of a randomized, vehicle-controlled study. Allergy. 2010 Dec;65(12):1594-9. doi: 10.1111/j.1398-9995.2010.02417.x. Epub 2010 Sep 7. PMID 21039597